CLINICAL TRIAL: NCT06735729
Title: Attitudes and Technical Maneuvers Regarding Enterostomy Management and Stoma Creation Among Surgeons: a Cross-sectional Study
Brief Title: Attitudes and Technical Maneuvers Regarding Enterostomy Management and Stoma Creation Among Surgeons
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lin Wang, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute
Other Study IDs: COCG-00
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Neoplasms; Colorectal Surgery
Keywords: surgeon attitude; surgical procedure; stoma; enterostomy; colorectal cancer; cross-sectional study
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- surgeons involved in stoma: All the surgeons were coming from either general surgery, gastrointestinal surgery, surgical oncology, emergency, and other departments involved stoma creation. their concepts and attitudes regarding to enterostomy management were investigated by a electronic questionnaire which comprised of five parts: personnel qualification and training, attitude toward stoma-related complications, preoperative siting, process of acquiring ostomy-related surgical skills, and awareness and adoption of relevant techniques (37 items in total).

SUMMARY:
This study was aiming to investigate Chinese surgeons' attitudes toward and technical preferences for stoma creation.

DETAILED DESCRIPTION:
The survey comprised five parts: personnel qualification and training, attitude toward stoma-related complications, preoperative siting, process of acquiring ostomy-related surgical skills, and awareness and adoption of relevant techniques (37 items in total). The questionnaire was distributed to Chinese hospitals by Sojump, a professional online platform. Finally, about 401 surgeons had responded including 188 hospitals of different grades across 26 provinces or municipalities directly under the Central Government.

ELIGIBILITY:
Inclusion Criteria: General or gastrointestinal surgeons involved in general surgery, gastrointestinal surgery, surgical oncology, emergency, and others involved in managing enterostomies who had completed their degree and were licensed, or at least resident surgeons were included.

-

Exclusion Criteria: Surgeons who did not provide consent to participate in this study were excluded.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the surgeons were coming from either general surgery, gastrointestinal surgery, surgical oncology, emergency, and other departments involved stoma creation. their concepts and attitudes regarding to enterostomy management were investigated by a electronic questionnaire which comprised of five parts: personnel qualification and training, attitude toward stoma-related complications, preoperative siting, process of acquiring ostomy-related surgical skills, and awareness and adoption of relevant techniques (37 items in total).
  At the end of the study, a total of 401 participants participated including 188 hospitals of different grades across 26 provinces or municipalities directly under the Central Government.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
attitude, technical preferences | 1 month
  surgeons' attitude and technical preferences information was collecting by the 37 items on the questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No